CLINICAL TRIAL: NCT05121142
Title: Pharmacokinetics and Pharmacodynamic Study of Ruxolitinib for the Management of Acute and Chronic Graft Versus Host Disease
Brief Title: Study of Ruxolitinib for Acute and Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0167
Record Dates: First submitted 2021-09-01; First posted 2021-11-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Acute-graft-versus-host Disease; Chronic Graft-versus-host-disease; Solid Organ Transplant
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Existing patients with chronic GVHD (No Intervention): Participants with established diagnosis of chronic GVHD and currently on treatment with ruxolitinib for chronic GVHD for at least 3 weeks. Participants in this arm are receiving ruxolitinib clinically and will not receive ruxolitinib as part of this research study.
- Arm 2: Acute GVHD ages 0-<12 years (Experimental): Participants with acute GVHD will receive ruxolitinib on this arm.
  Interventions: Drug: Ruxolitinib
- Arm 3: New onset chronic GVHD ages 0-≤18 years (Experimental): Participants with new onset chronic GVHD will receive ruxolitinib on this arm.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib will be given by mouth or enteral tube (if applicable).
  Arms: Arm 2: Acute GVHD ages 0-<12 years; Arm 3: New onset chronic GVHD ages 0-≤18 years

SUMMARY:
While hematopoietic stem cell transplant (HSCT) is an effective therapy, graft versus host disease (GVHD) is the most significant complication after HSCT. Both acute GVHD and chronic GVHD are leading causes of non-relapse morbidity and mortality. Patients with solid organ transplants may participate in this study as well because these patients occasionally develop acute GVHD, which is biologically similar to acute GVHD after an HSCT.

Acute graft versus host disease usually occurs within the first 100 days of transplant and can involve the skin, gut, or liver. Chronic graft versus host disease usually occurs after the first 100 days of transplant and can involve skin, eyes, mouth, joints, liver, intestines commonly. These two diseases are different, but both happen due to the imbalance of the donor immune system in the host.

The purpose of this research is to learn more about ruxolitinib as a treatment for both acute and chronic GVHD. Specifically, the investigators would like to learn more about the pharmacokinetics (PK - the process of absorption, distribution, metabolism, and elimination from the body - meaning how the drug moves through the body) and the pharmacodynamics (PD - the body's biological response to the drug) of ruxolitinib.

ELIGIBILITY:
ARM 1

Inclusion Criteria:

* Established diagnosis of chronic GVHD (all grades eligible)
* Currently on treatment with ruxolitinib for chronic GVHD for a minimum of 3 weeks
* No changes in doses of ruxolitinib or concurrent azoles (if present) one week prior to obtaining ruxolitinib levels
* Ages eligible for enrollment (0-≤18 years at time of enrollment)

Exclusion Criteria:

* Clinical presentation resembling overlap syndrome with both acute and chronic GVHD features

ARM 2

Inclusion Criteria:

* Ages <12 years status post allogeneic hematopoietic stem cell transplant or solid organ transplant
* Any underlying diagnoses, preparative regimen, stem cell source or acute GVHD prophylaxis are eligible
* Diagnosis of acute GVHD which is refractory to steroids (defined as lack of improvement to 2 mg/kg/day of methylprednisolone or bioequivalent oral steroids, for 7 days or progression of acute GVHD within 72 hours at 2 mg/kg/day of Methylprednisolone or bioequivalent oral doses)
* Able to take enteral medications
* Clinically diagnosed Grades II to IV acute GVHD as per modified Glucksberg criteria occurring after allogeneic HSCT requiring systemic immune suppressive therapy. Biopsy of involved organs with acute GVHD is encouraged but not required for study enrollment.
* Blood counts at decision to initiate ruxolitinib: absolute neutrophil count (ANC) > 1000/mm3* AND platelets ≥ 20,000/mm3 (*Use of growth factor supplementation and transfusion support is allowed to achieve these above defined hematological parameters)
* Estimated GFR by cystatin C of >30 mL/min
* Prior systemic treatments for acute GVHD are allowed. Once ruxolitinib is initiated, no further doses of these agents will be allowed.
* Calcineurin inhibitors are allowed throughout the duration of study and may be discontinued per treating physician discretion. Additionally dose adjustments to maintain target blood levels of calcineurin inhibitors may proceed per routine clinical practice.

Exclusion Criteria:

* Clinical presentation resembling de novo chronic GVHD or GVHD overlap syndrome with both acute and chronic GVHD features
* Presence of an active uncontrolled infection including significant bacterial, fungal, viral or parasitic infection requiring treatment. Infections are considered controlled if appropriate therapy has been instituted and no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Evidence of uncontrolled viral reactivation (Adenovirus, CMV, EBV, BK virus). If patients are on appropriate antiviral therapy or have received virus specific T-cells (either donor derived or third-party) then the viral reactivation is not considered uncontrolled.
* Presence of relapsed primary malignancy.

ARM 3

Inclusion Criteria:

* 0-≤18 years of age are eligible
* Any underlying diagnosis, preparative regimen, stem cell source or prior acute GVHD prophylaxis are eligible
* Diagnosis of chronic GVHD as per 2014 NIH consensus criteria (any organ involvement is eligible)
* Any GVHD global severity is eligible
* Patients may have received methylprednisolone or oral bioequivalent steroids at a dose of 1 mg/kg/day (or greater) for up to 28 days prior to enrollment but may be enrolled anytime between diagnosis of chronic GVHD and day 28 of systemic steroids
* Concurrent local therapies ( including but not limited to topical steroids, topical calcipotriene, ocular drops such as restasis, autologous serum eye drops, artificial tears, triamcinolone ointment for vulvar GVHD, Fluticasone Azithromycin and Singulair) are allowed at anytime while on ruxolitinib . Additional therapies may also be considered with PI review and approval
* As children may not meet criteria for lung GVHD due to inability to perform PFTs we will establish the diagnosis of lung GVHD for children as defined by any of the following criteria listed below. However, the participants do not need to have lung involvement to be eligible to receive ruxolitinib.

  1. >10% decrease in FEV1 or FVC from baseline or 25% of FEF 25-75
  2. Active GVHD in another organ system + pulmonary symptoms (Tachypnea without wheezing, new oxygen requirement, cough)
  3. Increased R5 by 50% by Impulse oscillometry
  4. Air trapping on high resolution CT scan, small airway thickening, or bronchiectasis in the absence of infection
* Negative urine or serum pregnancy test for females of childbearing age
* Estimated GFR by cystatin C > 30 mL/min
* Able to take enteral medications

Exclusion Criteria:

* Clinical presentation resembling overlap syndrome with both acute and chronic GVHD features
* Presence of an active uncontrolled infection including significant bacterial, fungal, viral or parasitic infection requiring treatment. Infections are considered controlled if appropriate therapy has been instituted and no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Evidence of uncontrolled viral reactivation (Adenovirus, CMV, EBV, BK virus). If patients are on appropriate antiviral therapy or have received virus specific T-cells (either donor derived or third-party) then the viral reactivation is not considered uncontrolled.
* Presence of relapsed primary malignancy.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2023-05-13 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
Cmax of ruxolitinib in existing patients with chronic GVHD (Arm 1) | 1 week
  Maximum Plasma Concentration of ruxolitinib
Cmax of ruxolitinib in patients with acute GVHD (Arm 2) | 30 days
  Maximum Plasma Concentration of ruxolitinib
Cmax of ruxolitinib in patients with new onset chronic GVHD (Arm 3) | 6 months
  Maximum Plasma Concentration of ruxolitinib
To measure phosphorylation of STAT5 on lymphocytes as a functional measure of JAK inhibition (Arms 1, 2, and 3) | Approximately 2 hours after the ruxolitinib dose
  A blood sample will be collected at the specified time point and pharmacodynamics will be measured by PSTAT5

SECONDARY OUTCOMES:
Number of participants with overall survival (Arm 3) | 6 months after ruxolitinib initiation
Number of participants with complete response to ruxolitinib (Arm 2) | 30 days after ruxolitinib initiation
  Complete response is defined as resolution of acute GVHD
Number of participants with partial response to ruxolitinib (Arm 2) | 30 days after ruxolitinib initiation
  Partial response is defined as improvement in stage of at least one organ involved in acute GVHD without worsening in additional organs
Number of participants with no response to ruxolitinib (Arm 2) | 30 days after ruxolitinib initiation
  No response is defined as lack of improvement or worsening of acute GVHD
Number of participants with response to ruxolitinib (Arm 3) | 6 months after ruxolitinib initiation
  Response is defined as resolution of chronic GVHD in at least one organ without worsening in additional organs
Number of participants with relapse free survival at 6 months (Arm 3) | 6 months after ruxolitinib initiation
Number of participants with relapse free survival at 6 months (Arm 1) | 6 months after ruxolitinib initiation
  Relapse free survival at 6 months for participants on Arm 1 only if participant has been on ruxolitinib clinically for 6 months
Incidence of infections (Arm 1) | through study completion, average of 7 days
  Infections defined as bacterial, parasitic, fungal, new viral reactivation or disease
Incidence of infections (Arm 2) | 30 days after ruxolitinib initiation
  Infections defined as bacterial, parasitic, fungal, new viral reactivation or disease
Incidence of infections (Arm 3) | 6 months after ruxolitinib initiation
  Infections defined as bacterial, parasitic, fungal, new viral reactivation or disease
Incidence of known side effects (Arm 1) | through study completion, average of 7 days
  Known side effects are defined as the side effects included in the Investigator's Brochure
Incidence of known side effects (Arm 2) | 30 days after ruxolitinib initiation
  Known side effects are defined as the side effects included in the Investigator's Brochure
Incidence of known side effects (Arm 3) | 6 months after ruxolitinib initiation
  Known side effects are defined as the side effects included in the Investigator's Brochure
Incidence of unknown side effects (Arm 1) | through study completion, average of 7 days
  Unknown side effects are defined as the side effects not included in the Investigator's Brochure
Incidence of unknown side effects (Arm 2) | 30 days after ruxolitinib initiation
  Unknown side effects are defined as the side effects not included in the Investigator's Brochure
Incidence of unknown side effects (Arm 3) | 6 months after ruxolitinib initiation
  Unknown side effects are defined as the side effects not included in the Investigator's Brochure
Number of participants who were weaned off steroids (Arm 2) | 30 days after ruxolitinib initiation
  Participants will be considered weaned off steroids if the steroid dose has been decreased
Number of participants who were weaned off steroids (Arm 3) | 6 months after ruxolitinib initiation
  Participants will be considered weaned off steroids if the steroid dose has been decreased

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Khandelwal, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No